CLINICAL TRIAL: NCT06463470
Title: Cognitive Behavioural Therapy for Avoidant/Restrictive Food Intake Disorder (CBT-AR): An Evaluation of the Feasibility, Acceptability and Effectiveness in Individuals Aged 12 to 25 Years
Brief Title: Cognitive Behavioural Therapy for Avoidant/Restrictive Food Intake Disorder (CBT-AR)
Acronym: CBT-AR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orygen (Other)
Collaborators: University of Melbourne (Other); Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORY-P02-24-04
Record Dates: First submitted 2024-05-30; First posted 2024-06-17 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Avoidant/Restrictive Food Intake Disorder (ARFID)
Keywords: Mental Health; Eating Disorders
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Psychological Well-Being; Feeding and Eating Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Non-randomised evaluation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Behavioural Therapy for Avoidant/Restrictive Food Intake Disorder (CBT-AR) (Experimental): This therapy involves four stages.
  * Stage 1 -Psychoeducation: This is covered in 2-4 sessions and involves explaining what ARFID is, educating patients and carers on food groups, nutrition and how to develop a balanced diet. Work is also done to increase eating volume for those who are underweight.
  * Stage 2 -Treatment planning: This is covered in 2 sessions and involves matching the individuals needs to the correct exposure approach (examples provided in stage 3).
  * Stage 3 -Graded exposure is covered for between 12 and 22 sessions (depending on the patient's needs) and describes slowly introducing more variety and volume of foods into the patient's diet.
  * Stage 4 -Relapse prevention: This is covered in 2 sessions. In these sessions, individuals are taught to recognise triggers and indicators of relapse. They are then able to go back to the materials provided in treatment to guide their management of these relapsing thoughts/behaviours.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Avoidant/Restrictive Food Intake Disorder (CBT-AR)

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Avoidant/Restrictive Food Intake Disorder (CBT-AR) — CBT-AR describes an adaption of cognitive behavioural therapy for use with individuals diagnosed with Avoidant/Restrictive Food Intake Disorder (ARFID).

SUMMARY:
CBT-AR describes an adaption of cognitive behavioural therapy for use with individuals diagnosed with Avoidant/Restrictive Food Intake Disorder (ARFID). The purpose of this evaluation is to determine the feasibility, acceptability and effectiveness of this treatment.

It is hypothesised that this treatment will be feasible and acceptable to clinicians, carers and patients and will be effective in reducing symptoms of ARFID for patients.

DETAILED DESCRIPTION:
CBT-AR describes an adaption of cognitive behavioural therapy that is appropriate for use with individuals diagnosed with Avoidant/Restrictive Food Intake Disorder (ARFID). This therapy will be delivered by trained clinicians (e.g. psychologists, mental health nurses) and involves weekly sessions for 18-30 sessions (up to 30 sessions for underweight patients). This therapy will be delivered face-to-face whenever possible. If required (participant not able to travel for a session etc.) online or telephone sessions will be conducted.

This therapy involves four stages as described below.

* Stage 1 - Psychoeducation: This is covered in 2-4 sessions and involves explaining what ARFID is, educating patients and carers on food groups, nutrition and how to develop a balanced diet. Work is also done to increase eating volume for those who are underweight.
* Stage 2 - Treatment planning: This is covered in 2 sessions and involves matching the individuals needs to the correct exposure approach (examples provided in stage 3).
* Stage 3 - Graded exposure is covered for between 12 and 22 sessions (depending on the patient's needs) and describes slowly introducing more variety and volume of foods into the patient's diet. For those patients who are uncomfortable with strong tastes and textures, graded exposure might involve eating very small amounts of new foods during which time they are encouraged to describe the look, feel and taste of the food using neutral words to reduce a negative response. If they have a fear of choking, they might start by talking about that fear, followed by watching a video of someone choking and recovering, then they might eat a very small amount of food to reduce the risk of choking, followed by increases in portions over time.
* Stage 4 - Relapse prevention: This is covered in 2 sessions. In these sessions, individuals are taught to recognise triggers and indicators of relapse. They are then able to go back to the materials provided in treatment to guide their management of these relapsing thoughts/behaviours.

Clinicians will collect data on adherence weekly. A measure of patient, parent/guardian and clinician satisfaction will be collected at the end of stage 4.

Parents/guardians of individuals <16yrs, or parents/guardians of patients who are underweight and living at home irrespective of age are involved in therapy through attending psychoeducation sessions and supporting the completion of homework.

ELIGIBILITY:
Inclusion Criteria:

* Current primary diagnosis of ARFID according to DSM-5 criteria as determined by the treating team (the eating disorders Orygen Specialist Program
* Presenting for treatment in the eating disorders Orygen Specialist Program
* If <16yo, or >16 but underweight (BMI <18.5) and living with their parents/guardian, a parent/guardian should be involved in the treatment.

Exclusion Criteria:

* Current tube feeding
* Inappropriateness for CBT-AR as determined by the clinicians (e.g. if there are more urgent issues to first manage such as high suicidal ideation, if participants do not have adequate comprehension capability, etc)

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-06-27 (Estimated); Study Completion 2027-06-27 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Upon conclusion of the study (week 18-30)
  Feasibility will be determined based on whether patients attended sessions. This information will be collected weekly.
  Clinicians will also record if a patient drops out of therapy and why (if known)
Acceptability: CTS | The CTS will be completed upon conclusion of the study (week 18-30)
  This outcome will be measured using 'The Compliance to Treatment Schedule' (CTS).
Acceptability: CSQ | The CSQ will be completed upon conclusion of the study (week 18-30)
  This outcome will be measured using the 'Client Satisfaction Questionnaire' (CSQ). Scores range from 8-32, with higher scores indicative of greater satisfaction.
Acceptability: Adverse events | Adverse events will be collected weekly between baseline and the conclusion of the study (week 18-30)
  This outcome will be measured using recordings of adverse events. Adverse events will be monitored weekly. Participants will be asked open-ended questions to determine whether they have experienced an adverse event in the past week. If an adverse event is elicited, in addition to describing the event and associated treatments, clinicians will ask questions to determine the severity and seriousness of the event, the likelihood that it is related to CBT-AR, and the outcome of the event. Examples of possible events might include vomiting or an allergic reaction to food in session or heightened anxiety around eating between sessions.
Acceptability: Qualitative Feedback | Qualitative feedback will be collected at the conclusion of the study (end of stage 4, week 20-30)
  This outcome will be measured using recordings of qualitative feedback. Qualitatively, clinicians are given an open text box and invited to enter any comments they might have including comments relating to the acceptability of the treatment.
Effectiveness: PARDI-AR-Q | The PARDI-AR-Q will be assessed at baseline, and at the conclusion of stages 2 (week 4-6) and 3 (week 18-28) and at conclusion of the study (week 18-30)
  This outcome will be measured using the Pica, ARFID, and Rumination Disorder Interview - ARFID Questionnaire (PARDI-AR-Q). Scores range from 0-6 for each subscale of severity of impact, sensory based avoidance, lack of interest, and concern about aversive consequences, with higher scores indicating greater severity.
Effectiveness: FNS | The FNS will be assessed at baseline and weekly and upon conclusion of the study (week 18-30)
  This outcome will be measured using the Food Neophobia Scale (FNS). Scores range from 0-42 on the shortened FNS, with higher scores indicative of greater food neophobia.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | BMI will be assessed at baseline and weekly and upon conclusion of the study (week 18-30)
  Calculated using weight and height Weight will be measured using digital scales and height measured using stadiometer
Distress | The DASS-Y will be assessed at baseline and at the conclusion of stages 2 and 3 and at conclusion of the study (week 18-30)
  Depression, Anxiety, Stress Scale for Youth (DASS-Y). Scores range from 0-42 on each subscale of depression, anxiety and stress, with higher scores indicating greater severity.
Quality of life (QoL) | The ReQol will be assessed at baseline and at the conclusion of stages 2 and 3 and at conclusion of the study (week 18-30)
  Recovering Quality of Life Questionnaire (ReQol). Scores range from 0-40 with higher scores indicating higher quality of life.
Quality of the relationship between clinician and patient | This will be measured upon conclusion of the study (week 18-30)
  Working Alliance Inventory - Short Revised (WAI-SR). Scores range from 4-20 on each of the subscales of agreement of tasks, goals and bond, with higher scores indicative of stronger therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Phillipou, Principal Investigator — Orygen
Locations (2):
- Australia (2):
  - Orygen Youth Health - Sunshine - Sunshine, Melbourne, Victoria
  - Orygen Youth Health - Parkville - Parkville, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No